CLINICAL TRIAL: NCT01219738
Title: Acute Airway Vascular Smooth Muscle Effects of Inhaled Budesonide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Eliana Mendes, University of Miami, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 20071068; IRUSBUPF0002 (Other: Sponsor)
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
Keywords: Asthma, airway blood flow, budesonide, glucocorticosteroid.
MeSH Terms: conditions — Asthma | interventions — Budesonide; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- budesonide 360ug (Experimental): asthmatic subject received different doses of inhaled budesonide in random other
  Interventions: Drug: Budesonide 360ug
- budesonide 720ug (Experimental): asthmatic subject received different doses of inhaled budesonide in random other
  Interventions: Drug: Budesonide 720ug
- budesonide 1440ug (Experimental): asthmatic subject received different doses of inhaled budesonide in random other
  Interventions: Drug: Budesonide 1440ug
- placebo (Placebo Comparator): asthmatic subject received inhaled placebo
  Interventions: Drug: Budesonide720ug 4 times
- Budesonide720ug 4 times (Experimental): asthmatic subject received 720ug of inhaled budesonide 4 times separated by 30 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide 360ug — A single inhaled dose of 360ug budesonide from a DPI.
  Other Names: Pulmicort Flexhaler
  Arms: budesonide 360ug
Drug: Budesonide 720ug — A single inhaled dose of 720ug budesonide from a DPI.
  Other Names: Pulmicort Flexhaler
  Arms: budesonide 720ug
Drug: Budesonide 1440ug — A single dose of 1440ug of the budesonide from DPI.
  Other Names: Pulmicort Flexhaler
  Arms: budesonide 1440ug
Drug: Budesonide720ug 4 times — 720ug of budesonide will be inhaled by the subjects 4 times, separated by 30 minutes.
  Other Names: Pulmicort Flexhaler
  Arms: placebo
Drug: Placebo — A single inhaled dose of placebo from a DPI.
  Other Names: sugar pill
  Arms: Budesonide720ug 4 times

SUMMARY:
Glucocorticosteroids recently have been shown to have non-genomic actions that are plasma membrane-mediated and do not require gene transcription and translation. One of these non-genomic effects is the inhibition of adrenergic agonist transport into airway vascular smooth muscle cells with an increase of adrenergic agonist concentrations at adrenergic receptor sites and enhance the physiological effects of endogenous adrenergic agonists (e.g. locally released norepinephrine from noradrenergic neurons) or exogenous adrenergic agonists (e.g. inhaled beta-adrenergic agonists).

DETAILED DESCRIPTION:
Inhaled glucocorticosteroids typically are not recommended for the treatment of acute asthma attacks. This practice is based on the fact that glucocorticosteroids by themselves do not cause rapid bronchodilation. However, the acute inhibition of adrenergic agonist disposal by the non-genomic action of glucocorticosteroids could lead to bronchial vasoconstriction by locally released norepinephrine thereby decongesting the airway wall, and potentiate the bronchodilator effect of a concomitantly administered beta-adrenergic agonist through the same mechanism. The purpose of this study is to assess the vasoconstrictive effects of single and repetitive high-dose budesonide inhalations in moderate to severe asthmatics who use inhaled glucocorticosteroids regularly. As a secondary endpoint, airway inflammation and airway function will also be measured with the expectation that acute improvements in airflow might be detectable as a result of airway decongestion, notably in subjects with moderately severe asthma who have lower baseline lung function.

ELIGIBILITY:
Inclusion Criteria:

Twenty lifetime nonsmokers moderate or severe asthmatics; FEV1≥50 of predicted on the screening day

Exclusion Criteria:

Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women; Cardiovascular disease and/or use of cardiovascular medication; Subjects with known beta-adrenergic agonist or glucocorticosteroid intolerance; Acute respiratory infection and or acute exacerbation of asthma within four weeks prior to the study; Use of systemic glucocorticosteroids within 4 weeks prior to the study; Daily ICS dose (fluticasone or budesonide) > 500ug; Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliana Mendes, MD, Principal Investigator — University of Miami
Locations (1):
- Pulmonary Human Research Laboratory, University of Miami, Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Horvath G, Sutto Z, Torbati A, Conner GE, Salathe M, Wanner A. Norepinephrine transport by the extraneuronal monoamine transporter in human bronchial arterial smooth muscle cells. Am J Physiol Lung Cell Mol Physiol. 2003 Oct;285(4):L829-37. doi: 10.1152/ajplung.00054.2003. Epub 2003 Jun 13. PMID 12807698
- [Background] Horvath G, Lieb T, Conner GE, Salathe M, Wanner A. Steroid sensitivity of norepinephrine uptake by human bronchial arterial and rabbit aortic smooth muscle cells. Am J Respir Cell Mol Biol. 2001 Oct;25(4):500-6. doi: 10.1165/ajrcmb.25.4.4559. PMID 11694456
- [Background] Mendes ES, Pereira A, Danta I, Duncan RC, Wanner A. Comparative bronchial vasoconstrictive efficacy of inhaled glucocorticosteroids. Eur Respir J. 2003 Jun;21(6):989-93. doi: 10.1183/09031936.03.00072402. PMID 12797493
- [Background] Brieva JL, Danta I, Wanner A. Effect of an inhaled glucocorticosteroid on airway mucosal blood flow in mild asthma. Am J Respir Crit Care Med. 2000 Jan;161(1):293-6. doi: 10.1164/ajrccm.161.1.9905068. PMID 10619834
- [Derived] Mendes ES, Rebolledo P, Campos M, Wanner A. Immediate antiinflammatory effects of inhaled budesonide in patients with asthma. Ann Am Thorac Soc. 2014 Jun;11(5):706-11. doi: 10.1513/AnnalsATS.201307-220OC. PMID 24735128

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: asthmatic subject received different doses of inhaled budesonide
  Budesonide: A single inhaled dose of 360ug budesonide from a DPI.
  Budesonide: A single inhaled dose of 720ug budesonide from a DPI.
  Budesonide: A single dose of 1440ug of the budesonide from DPI.
  Budesonide: 720ug of budesonide will be inhaled by the subjects 4 times, separated by 30 minutes.
  Placebo: A single inhaled dose of placebo from a DPI.
Period: Overall Study
Arm/Group | All Study Participants
Started | 20
Budesonide 360 | 20
Budesonide 720 | 20
Budesonide 1440 | 20
Budesonide 720- 4 Times | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Asthma: asthmatic subject received different doses of inhaled budesonide
  Budesonide: A single inhaled dose of 360ug budesonide from a DPI.
  Budesonide: A single inhaled dose of 720ug budesonide from a DPI.
  Budesonide: A single dose of 1440ug of the budesonide from DPI.
  Budesonide: 720ug of budesonide will be inhaled by the subjects 4 times, separated by 30 minutes.
  Placebo: A single inhaled dose of placebo from a DPI.
Arm/Group | Asthma
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 43 [22 to 66]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20
Airway blood flow [Mean (Standard Deviation); unit: μl/min/ml] | 52.3 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Airway Blood Flow (Qaw)
Description: Qaw will be measured before and up to 6 hours after a single inhaled dose of 360ug, 720ug, and 1440ug budesonide or placebo from a DPI, using a double-blinded randomized design on different days.
Time Frame: participants will be followed for 6 hours after budesonide dose
Measure: Mean (Standard Error); unit: percentage of change from baseline
Groups:
- Budesonide 360ug: Budesonide: A single inhaled dose of 360ug budesonide from a DPI.
- Budesonide 720ug: Budesonide: A single inhaled dose of 720ug budesonide from a DPI.
- Budesonide 1440ug: Budesonide: A single dose of 1440ug of the budesonide from DPI.
- Budesonide 720ug 4 Times: Budesonide: 720ug of budesonide will be inhaled by the subjects 4 times, separated by 30 minutes.
Arm/Group | Budesonide 360ug | Budesonide 720ug | Budesonide 1440ug | Budesonide 720ug 4 Times | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 20
percentage of change from baseline | 22.3 (2.1) | 29.4 (2.7) | 34.1 (2.5) | 28.2 (1.9) | 5.1 (2.4)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 will be measured before and up to 6 hours after a single inhaled dose of 360ug, 720ug, and 1440ug budesonide or placebo from a DPI, using a double-blinded randomized design on different days.
Time Frame: participant will be followed up to 6 hours after budesonide dose
Measure: Mean (Standard Error); unit: percentage of change from baseline
Groups:
- Budesonide 360 ug: Budesonide: A single inhaled dose of 360ug budesonide from a DPI.
- Budesonide 720 ug: Budesonide: A single inhaled dose of 720ug budesonide from a DPI.
- Budesonide 1440 ug: Budesonide: A single inhaled dose of 1440ug budesonide from a DPI.
- 720ug of Budesonide 4 Times: Budesonide: 720ug of budesonide will be inhaled by the subjects 4 times, separated by 30 minutes.
Arm/Group | Budesonide 360 ug | Budesonide 720 ug | Budesonide 1440 ug | 720ug of Budesonide 4 Times | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 18 | 20
percentage of change from baseline | 0.1 (0.6) | 3.2 (1.9) | 1.6 (1.8) | 3.2 (2.4) | 0.8 (2.8)

ADVERSE EVENTS:
Time Frame: overall study, up to six hour after each dose.
Groups:
- All Study Participants: Budesonide:was given in different doses
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes